CLINICAL TRIAL: NCT04977128
Title: Safety Study of 89Zr-labeled KN035 PET Imaging in Patients With PD-L1 Positive Solid Tumors
Brief Title: 89Zr-labeled KN035 PET Imaging in Patients With PD-L1 Positive Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wuxi 4 PDL1 202106
Record Dates: First submitted 2021-07-06; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：89Zr-KN035 injection (Experimental): Patients will receive a tracer (10 mg, IV) dose of Zr-89 (2-3mCi) labelled KN035 (89Zr- KN035)
  Interventions: Drug: 89Zr-KN035

INTERVENTIONS:
Drug: 89Zr-KN035 — Patients will receive a tracer (10 mg, IV) dose of Zr-89 (2-3mCi) labelled KN035 (89Zr- KN035)

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 89Zr-labeled KN035 (89Zr-KN035) PET Imaging in patients with PD-L1 positive solid tumors.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Patients will receive an injection of 89Zr-KN035 and will undergo PET/CT scanning to determine uptake of 89Zr-KN035 in tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age 18-75, male or female;
3. Patients diagnosed with solid tumors confirmed by histopathology or cytology;
4. At least one measurable solid lesion has been examined by 18F-FDG PET/CT (RECIST1.1 standard);
5. Patients with biopsy-proven PD-L1 positive;
6. ECOG score ≤ 0~1; Life expectancy of at least 3 months;
7. Women of childbearing age are required to receive serum pregnancy tests, and only those who have a negative pregnancy test for eligible subjects.

Exclusion Criteria:

1. Currently or within the first 28 days before the first dose to participate in another therapeutic clinical trial. If participating in a non-interventional clinical trial, it is not be excluded;
2. Patients with systemic or locally severe infections (CTCAE ≥ 2);
3. Patients with allergies or allergies to any component of the imaging agent or antibody;
4. Patients who cannot undergo PET/CT imaging;
5. Intolerance of intravenous administration, as well as difficulties in venous blood collection (If having the medical history of fainting during acupuncture, and blood phobia);
6. Symptomatic congestive heart failure (NYHA class II-IV) or symptomatic or poorly controlled arrhythmia;
7. Patients have significant QT/QTC interval prolongation during the screening period;
8. Received anti-tumor therapy (including but not limited to chemotherapy, radiotherapy, biological therapy) within 4 weeks prior to first dose;
9. Patents have not recovered to CTCAE grade 0 or 1 from the adverse events due to cancer therapeutics administered;
10. Patients need to receive other anti-tumor treatments during the trial period；
11. Previously received CD137 agonist or immune checkpoint blocking therapy;
12. Patients with diabetes who have a fasting blood glucose greater than 10 mmol/L;
13. HIV antibody positive, active hepatitis B/C, and TB positive;
14. Patients are regular users (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol);
15. Patients with symptomatic ascites, pleural effusion, or hydropericardium;
16. Pregnant or lactating women, or planning to become pregnant or have children during this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of 89Zr-KN035 in PD-L1 positive solid tumor patients | 1 year
  Safety will be assessed by evaluation of incidence of adverse events

SECONDARY OUTCOMES:
Biodistribution of 89Zr-KN035 | 1 year
  The biodistribution of the tracer 89Zr-KN035 as assessed with 89Zr- KN035 PET scans.
Correlation 89Zr-KN035 uptake in tumor lesions and PD-L1 expression as determined by immunohistochemistry | 1 year
  Correlation 89Zr-KN035 uptake in tumor lesions and PD-L1 expression as determined by immunohistochemistry
Evaluation of immunotherapy efficacy | 1 year
  The correlation between the 89Zr-KN035 tumor uptake (Standardized uptake value SUV ) and response to therapy by performing 89Zr-KN035 scan before PD1 therapy， related to CT/MRI response according to RECIST1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi No. 4 People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided